CLINICAL TRIAL: NCT05823701
Title: A Phase 2 Study of Chidamide, Azacitidine Combined With GM Regimen for Patients With Relapsed and Refractory DLBCL
Brief Title: Chidamide, Azacitidine Combined With GM Regimen for Relapsed and Refractory DLBCL Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jinzm003
Record Dates: First submitted 2023-02-27; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2022-08

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Azacitidine; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide, Azacitidine Combined With GM(CAGM) Regimen (Experimental): R/R DLBCL patients were treated with 2 cycles of CAGM regimen including chidamide, azacitidine, obinutuzumab and liposomal mitoxantrone followed by imaging examination. Patients achieved CR/PR were exposed to ASCT/CAR-T therapy or additional 4 cycles of CAGM regimen in patients ineligible for ASCT/CAR-T therapy; whereas, patients with SD/PD were withdrawn from this study.
  Interventions: Drug: Chidamide; Drug: Azacitidine; Biological: obinutuzumab; Drug: Liposomal mitoxantrone

INTERVENTIONS:
Drug: Chidamide — 20 mg (4 capsules), d1, d4, d8, d11 orally per cycle
  Other Names: Tucidinostat
Drug: Azacitidine — 100mg d1- d5 subcutaneous injection per cycle
  Other Names: AZA
Biological: obinutuzumab — 1000mg d4 intravenous infusion per cycle
  Other Names: Gazyva
Drug: Liposomal mitoxantrone — 20mg/m2 d5 intravenous infusion per cycle
  Other Names: PLM60

SUMMARY:
To evaluate the efficacy and safety of CAGM regimen in R/R DLBCL patients and to provide a safe and more effective approach for R/R DLBCL patients.

DETAILED DESCRIPTION:
The study will start with an initial 2 cycles of induction therapy with CAGM containing chidamide, azacitidine, obinutuzumab and mitoxantrone liposome, orelabrutinib and rituximab，following imaging examinations to evaluate response rates. For patients feasible to CAR-T/ASCT, sequential CAR-T/ASCT treatment was given. For patients who were unable to undergo CAR-T/ASCT, 4 cycles of CAGM immunochemotherapy were carried out. Efficacy and safety of CAGM regimen in R/R DLBCL will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. At least one measurable lesion，measurable lymph nodes or masses of at least 15 millimeter (mm).
3. Histopathologically confirmed DLBCL.
4. Diseases refractory to first-line treatment (including CD20 monoclonal antibody and anthracycline) or relapsed after the last treatment.
5. Life expectancy > 3 months.
6. Appropriate organ function: Cardiac function: cardiac ejection fraction ≥50%; Liver function: alanine aminotransferase and aspartate aminotransferase ≤3 times the upper limit of normal; Renal function: serum creatinine clearance ≥30 mL/min; Lung function: SPO2>91% without oxygen;
7. Adequate bone marrow reserve: Hemoglobin ≥8 g/dL; Platelet count ≥75×10^9/L; Absolute neutrophil value ≥1.0×10^9/L; Platelet count ≥50×10^9/L, absolute neutrophil value ≥0.75×10^9/L if there is bone marrow invasion.
8. The patient has the ability to understand and is willing to provide written informed consent.
9. Agreement to practice birth control from the time of enrollment until the follow-up period of the study.

Exclusion Criteria:

1. Severe liver and kidney dysfunction (alanine aminotransferase, bilirubin, creatinine > 3 times the upper limit of normal);
2. Structural heart disease, leading to clinical symptoms or abnormal cardiac function (NYHA ≥ grade 2);
3. Uncontrolled active infection;
4. Concurrent presence of other tumors requiring treatment or intervention;
5. Current or expected need for systemic corticosteroid therapy;
6. Pregnant or lactating women.
7. Other psychological conditions that prevent patients from participating in the research or signing the informed consent.
8. In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or does not meet the requirements for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate(ORR) | At the end of Cycle 2 (each cycle is 28 days)
  The rate of patients who achieved CR or PR after treatment by CAGM regimen
Complete response rate(CRR) | At the end of Cycle 2 (each cycle is 28 days)
  The rate of patients who achieved CR after treatment by CAGM regimen

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events, Treatment-Related Adverse Events and Serious Adverse Events | initiation of study drug until 30 days after last dose
  The safety and tolerability of the therapeutic regimen measured by the incidence of treatment-emergent adverse events, treatment-related adverse events and serious adverse events.
Progression-free survival(PFS) | Up to 24 months after the end of last patients' treatment.
  PFS will be assessed from the first CAGM given to date of progression, relapse, death or end of follow-up.
Overal survival(OS) | Up to 24 months after the end of last patients' treatment.
  OS will be assessed from the first CAGM given to date of death or end of follow-up.
Overall response rate(ORR) | At the end of Cycle 6 (each cycle is 28 days)
  The rate of patients who achieved CR or PR after treatment by CAGM regimen
Complete response rate(CRR) | At the end of Cycle 6 (each cycle is 28 days)
  The rate of patients who achieved CR after treatment by CAGM regimen

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China